CLINICAL TRIAL: NCT01704430
Title: GLutamine Enterally After carDiac Surgery for Inflammation Attenuation and ouTcOme impRovement (GLADIATOR): A Phase II Randomized, Blinded, Placebo-Controlled Trial
Brief Title: Glutamine to Improve Outcomes in Cardiac Surgery
Acronym: GLADIATOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MAZ_CVICU_001
Record Dates: First submitted 2012-08-22; First posted 2012-10-11 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Nosocomial Infection
Keywords: Cardiac surgery; Cardiac bypass; Intensive Care; Nosocomial infection; Glutamine; Randomized trial
MeSH Terms: conditions — Cross Infection | interventions — Glutamine; maltodextrin

STUDY DESIGN:
Intervention Model Description: Glutamine
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutamine (Experimental): Oral/enteral glutamine 0.5 g/kg satisfactory body weight per day (divided doses every 8 hours) starting 6 hours post-operatively
  Interventions: Dietary Supplement: Glutamine
- Maltodextrin (Placebo Comparator): Oral/enteral maltodextrin 0.5 g/kg satisfactory body weight per day (divided doses every 8 hours) starting 6 hours post-operatively
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Glutamine — Enteric L-Glutamine
  Other Names: L-Glutamine
  Arms: Glutamine
Dietary Supplement: Maltodextrin — Enteric Maltodextrin
  Arms: Maltodextrin

SUMMARY:
Patients undergoing heart surgery with a heart-lung machine (termed cardiopulmonary bypass) are at an increased risk of having abnormal "inflammation" in their body after surgery. Such inflammation can contribute to slower recovery from surgery, an increased risk of infection, an increased risk of damage to organs other than the heart, and a more complicated course.

Prior research has suggested that using an oral protein supplement made of glutamine (an essential amino acid normally found in your body) can reduce the risk of inflammation, infection and the length of stay in hospital in patients who have suffered major trauma or a burn injury. The investigators believe reducing such inflammation after heart surgery may help promote recovery and reduce the risk of adverse events and complications.

The purpose of this preliminary study is to see if oral glutamine supplementation after heart surgery is practical, and contributes to a reduction in inflammation. The oral glutamine proposed in this study is based on what has been previously studied and what is considered safe.

DETAILED DESCRIPTION:
Hypothesis: We believe that early post-operative administration of enteral glutamine following cardiac surgery with cardiopulmonary bypass (CPB) in high risk patients will reduce inflammation and nonscomial infections, reduce length of ventilator support, reduce need for vasoactive support, reduce secondary organ dysfunction, reduce length of hospital stay in the CVICU, and reduce mortality.

Objectives:

* To assess the feasibility of early glutamine supplementation
* To evaluate the safety profile of early glutamine supplementation
* To evaluate efficacy the impact of early glutamine on clinically important post-operative complications and outcomes, including: systemic inflammation, nosocomial infections, mortality, and health resource utilization

Methods: Study Design, Setting, and Patient Population: The proposed study is a Phase II, randomized, blinded, placebo-controlled trial. This trial will be performed in the Cardiovascular Surgical Intensive Care Unit (CVICU) of the Mazankowski Alberta Heart Institute (MAHI), Alberta Health Services. The proposed trial plans to enroll 100 consecutive eligible patients.

Inclusion:

* Consent (obtained pre-operatively)
* Adult - aged 18 years or older;
* Planned cardiac surgery with CPB;
* Elevated risk for post-operative morbidity, defined by a pre-operative European System for Operative Cardiac Risk Evaluation (EuroSCORE) > 6.
* Able to receive enteral nutrition through nasal/oral gastric or post-pyloric feeding tube.

Exclusion:

* Planned heart or lung transplantation
* Planned cardiac surgery without cardiopulmonary bypass;
* Peri-operative support with extracorporeal membrane oxygenation (ECMO) or left ventricular assist device (LVAD).

Study Protocol: Eligible patients will be identified during pre-operative assessment in the pre-operative clinic (PAC). All eligible patients or their surrogate decision-making/legal guardian will then be approached to obtain informed written consent.

Each consenting participant will be randomly allocated (1:1) to receive post-operative enteral glutamine or identical placebo. Investigators, surgeons, intensivists, bedside nurses and participants will remain blinded to study allocation.

Glutamine supplementation will be dosed at 0.5 g/kg satisfactory body weight (SBW)/day divided every 8 hours, starting 6 hours post-operatively and continued for 5 days. The dose of 0.5 g/kg SBW/day was effective in clinical studies using enteral glutamine in critically ill and/or burn injured and major trauma patients. The glutamine supplementation or placebo will be delivered via naso- or oro-gastric feeding tube after confirmation of placement by chest X-ray. For participants who are extubated prior to 5 days, enteral glutamine will be given by mouth for the duration of the 5 day period. Glutamine and placebo will be mixed in orange juice to maintain blinding.

ELIGIBILITY:
Inclusion Criteria:

* Consent (obtained pre-operatively)
* Adult - aged 18 years or older;
* Planned cardiovascular surgery with cardiopulmonary bypass;
* Increased risk for post-operative morbidity, defined by a pre-operative European System for Operative Cardiac Risk Evaluation (EuroSCORE) > 6;
* Able to receive enteral nutrition through nasal/oral gastric or post-pyloric feeding tube.

Exclusion Criteria:

* Planned heart or lung transplantation
* Planned cardiovascular surgery without cardiopulmonary bypass;
* Peri-operative support with extracorporeal membrane oxygenation (ECMO) or left ventricular assist device (LVAD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2016-06-21 (Actual); Study Completion 2016-06-21 (Actual)

PRIMARY OUTCOMES:
Proportion of Eligible Patients Providing Consent to Participate | Date of surgery until date of hospital discharge, an expected average of 2 weeks
  Assess the FEASIBILITY of the protocol to (i) achieve >75% consent rate in eligible patients

SECONDARY OUTCOMES:
Acute Kidney Injury | Date of surgery until date of hospital discharge, an expected average of 2 weeks
Duration of mechanical ventilation | Date of surgery until date of hospital discharge, an expected average of 2 weeks
Duration of vasoactive support | Date of surgery until date of hospital discharge, an expected average of 2 weeks
Blood transfusion | Date of surgery until date of hospital discharge, an expected average of 2 weeks
Organ Dysfunction Score | Date of surgery until date of hospital discharge, an expected average of 2 weeks
  Post-operative changes to the Sequential Organ Failure Assessment score
Adverse events | Date of surgery until date of hospital discharge, an expected average of 2 weeks
  Evaluate the SAFETY and ADVERSE EFFECTS of (i) enteral glutamine; and (ii) COMPLICATIONS from feeding tube placement, including: epistaxis, feeding tube malposition, pneumothorax, esophageal injury, gastric mucosal irritation, gastrointestinal bleeding, unplanned feeding tube removal, and need for feeding tube reinsertion
Systemic inflammation | Date of surgery until the end of planned study intervention, expected 5-days
  Systemic Inflammation/immunomodulation: We will evaluate for increases and changes in systemic inflammation stratified by study intervention. This will aid in providing proof-of-concept of the biologic plausibility of the study intervention. The investigators propose to evaluate serial measures of C-reactive protein (CRP), chemiluminescent endotoxin activity assay (EAA), and interleukin-6 (IL-6).
Nosocomial infection | Date of surgery until date of hospital discharge, an expected average of 2 weeks
  Nosocomial infections: The investigators will specifically examine for the following infections during the period of hospitalization after surgery: superficial and deep sternal wound infections; mediastinitis; saphenous vein graft harvest site wound infections; ventilator associated and hospital acquired pneumonia; urinary tract infections; bloodstream infections; catheter-related blood stream infections; and decubitus ulcers.
Proportion of Randomized Patients Achieving Protocol Adherence | 5-days (date of surgery until the end of planned study intervention)
  Obtain > 90% protocol adherence

OTHER OUTCOMES:
Mortality | From the Date of Surgery until Date of Death or 90-days, whichever occurs first
Duration of ICU stay | Date of surgery until date of hospital discharge, an expected average of 2 weeks
Duration of hospital stay | Date of surgery until date of hospital discharge, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sean Bagshaw, Principal Investigator — University of Alberta; Gurmeet Singh, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Mazankowski Alberta Heart Institute, University of Alberta, Edmonton, Alberta